CLINICAL TRIAL: NCT03094819
Title: PROTECT2: Diabetes Care - Eye Exam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Retinal Care Inc. (Industry)
Collaborators: Dean A. McGee Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 09-PLN-001
Record Dates: First submitted 2016-04-01; First posted 2017-03-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (No Intervention): Participants randomized to Group 1 will be the control group. They will be observed while they receive usual eye care without any study intervention.
- Financial Incentive (Experimental): Participants randomized to the Financial Incentive group will be offered a financial incentive in conjunction with their usual eye care. They will receive usual care and a $25 payment if they obtain a confirmed eye examination.
  Interventions: Behavioral: Financial Incentive
- Retinal Care DR (Experimental): Participants randomized to the Retinal Care DR Service group will receive: (1) point of care risk assessment for vision-threatening diabetic retinopathy, (2) retinal specialist interpretation of their risk assessment data, and (3) care coordination designed to improve the eye examination rate for patients with diabetes at increased risk for vision-threatening diabetic retinopathy.
  Interventions: Behavioral: Retinal Care DR

INTERVENTIONS:
Behavioral: Financial Incentive — Participants will receive usual care and a $25 payment if they obtain a confirmed eye examination.
  Arms: Financial Incentive
Behavioral: Retinal Care DR — Participants will receive: (1) point of care risk assessment for vision- threatening diabetic retinopathy, (2) retinal specialist interpretation of their risk assessment data, and (3) care coordination designed to improve the eye examination rate for patients with diabetes at increased risk for vision- threatening diabetic retinopathy.
  Arms: Retinal Care DR

SUMMARY:
The PROTECT2 pilot study is a single cohort prospective study to gather pilot data and finalize operational details of the main study.

The PROTECT2 main study is a prospective randomized controlled multi-center three group clinical trial. The primary endpoint is the percentage of participants in each study group obtaining a qualified eye examination within 12 months of their enrollment in the study.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the qualified eye examination rate in two groups of patients with diabetes receiving a new intervention, with the rate in a control group of patients with diabetes receiving usual care only.

Secondary objectives are to:

* Improve our understanding of the barriers to obtaining eye examinations;
* Evaluate the communication between eye care providers (ECP) and referring primary care providers (PCP), as determined by rates of follow-up reports sent and received;
* Characterize eye examinations provided to patients with diabetes;
* Explore the relationships between systemic variables known to affect the severity of diabetic retinopathy and the patient's risk of vision-threatening diabetic retinopathy.

Design and Primary Endpoint

* The pilot study is a single cohort prospective study to gather pilot data and finalize operational details of the main study.
* The main study is a prospective randomized controlled multi-center three group clinical trial. The primary endpoint is the percentage of participants in each study group obtaining a qualified eye examination within 12 months of their enrollment in the study.

Interventions and Duration

Eligible patients will be randomized to one of three groups in a 1:1:2 ratio.

* Group 1. Participants randomized to Group 1 will be the control group. They will be observed while they receive usual eye care without any study intervention.
* Financial Incentive. Participants randomized to the Financial Incentive group will be offered a financial incentive in conjunction with their usual eye care. They will receive usual care and a $25 payment if they obtain a confirmed eye examination.
* Retinal Care DR Service. Participants randomized to the Retinal Care DR Service group will receive: (1) point of care risk assessment for vision- threatening diabetic retinopathy, (2) retinal specialist interpretation of their risk assessment data, and (3) care coordination designed to improve the eye examination rate for patients with diabetes at increased risk for vision- threatening diabetic retinopathy.

All participants, regardless of their group, will be in the study for about one year.

Sample Size and Population Patients meeting the inclusion and exclusion criteria will be recruited at up to four (4) study sites until the sample size of 4,500 participants is enrolled. This includes up to 500 patients at each site in the pilot study, and weighted randomization in the main study to ensure enrollment of approximately 500 patients in the Retinal Care DR Service group at each site to evaluate the operational characteristics of the Retinal Care DR Service in populations representative of those anticipated in commercial use.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed diabetes using the criteria documented in the 2016 Physician Quality Reporting System (PQRS) Measure Specifications Manual for Claims and Registry Reporting of Individual Measures.
2. 18 through 75 years of age
3. Have a PCP appointment scheduled within 90 days of the date of medical record review.

Exclusion Criteria:

1. Patients not diagnosed with diabetes
2. History of photosensitive epilepsy
3. Inability or unwillingness of the participant to give verbal or written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2016-03-17 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualified eye examination rate | 12 months
  Percent of participants in each study group obtaining a qualified eye examination.

SECONDARY OUTCOMES:
PCP report rate | 12 months
  Percent of eye examinations with a follow-up report sent to the PCP.
PCP medical record rate | 12 months
  Percent of eye examinations with a follow-up report sent to the PCP, where the results of the follow-up report are documented in the PCP medical record.
Eye examination barriers | 12 months
  Descriptive analysis of barriers to obtaining an eye examination.
Increased risk group eye examination rate | 12 months
  Percent of participants at increased risk for vision-threatening diabetic retinopathy who are subsequently seen by an eye care provider.
Eye examination findings | 12 months
  Descriptive analysis of eye examination findings for participants at increased risk for vision-threatening diabetic retinopathy.
Eye examination components | 12 months
  Descriptive analysis of eye examination components for participants at increased risk for vision-threatening diabetic retinopathy.
Eye care costs | 12 months
  Numerical analysis of eye care costs using provider reported and claims data.
Risk correlations | 12 months
  Correlation analysis of systemic variables known to affect the severity of diabetic retinopathy and retinal specialist interpretation of participant's risk assessment data.
Participant perceptions | 12 months
  Descriptive analysis of participant perceptions of the Retinal Care DR Service.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Kingsley, MD, Principal Investigator — Dean McGee Eye Institute / University of Oklahoma Health Sciences Center
Locations (1):
- Dean McGee Eye Institute, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No